CLINICAL TRIAL: NCT05653830
Title: Multicenter, Retrospective-prospective, Observational Clinical Study of the Natural Course and Long-term Prognosis of Patients With Chronic Liver Disease
Brief Title: Observational Clinical Study of the Natural Course and Long-term Prognosis of Patients With Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Ankang Central Hospital (Other); 3201 Hospital in Hanzhong (Other); Weinan Central Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Tang-Du Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); General Hospital of Ningxia Medical University (Other); Lanzhou University Second Hospital (Other); First Affiliated Hospital of Lanzhou University (Unknown); The Fourth People's Hospital of Qinghai Province (Other); Yan'an University Affiliated Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-300
Record Dates: First submitted 2022-12-09; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-08

CONDITIONS: Chronic Liver Disease
Keywords: retrospective-prospective, observational clinical study of chronic liver disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 3 ml of serum was retained for prospective patient and stored frozen below -80 degrees
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients with chronic hepatitis B: Patients who meet the diagnostic criteria for chronic hepatitis B for long-term follow-up
- Patients with chronic hepatitis C: Patients who meet the diagnostic criteria for chronic hepatitis C for long-term follow-up
- Patients with chronic hepatitis D: Patients who meet the diagnostic criteria for chronic hepatitis D for long-term follow-up
- Patients with autoimmune liver disease（PBC\AIH\PSC）: Patients who meet the diagnostic criteria for autoimmune liver disease（PBC\AIH\PSC） for long-term follow-up
- Patients with NAFLD: Patients who meet the diagnostic criteria for NAFLD for long-term follow-up
- Patients with ALD: Patients who meet the diagnostic criteria for ALD for long-term follow-up

SUMMARY:
Chronic liver disease is a global public health problem. Without timely diagnosis and treatment, chronic liver disease can progress to hepatitis, liver fibrosis, and cirrhosis, while causing a variety of complications such as gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome, and liver cancer. Early detection and treatment can slow down the progression of chronic liver disease and reduce the burden of patients. This study intends to construct a retrospective-prospective cohort of patients with chronic liver disease by building a multicenter collaborative network to study the disease characteristics, progression patterns, clinical features, natural course and long-term prognosis of chronic liver disease of different etiologies.

DETAILED DESCRIPTION:
Different etiologies can lead to chronic liver disease, and common causes include non-alcoholic fatty liver disease (NAFLD), hepatitis B virus (HBV), hepatitis C virus (HCV), alcohol-related liver disease (ALD), primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC) and autoimmune hepatitis (AIH). In recent years, with the popularization of HBV vaccination and the advancement of drugs for the treatment of viral hepatitis, the incidence of cirrhosis has been curbed in many countries, but obesity, metabolic syndrome and alcohol abuse have led to an increase in the incidence of NAFLD and ALD recently. The large number of patients with cirrhosis causes loss of social workforce and depletion of medical resources, as well as increased family stress and reduced quality of life. As a result of that, cirrhosis remains a public health problem that cannot be ignored.

To better understand the natural course and clinical characteristics of chronic liver disease due to different etiologies, this study proposes to establish a multicenter, large sample, long-term follow-up cohort of patients with chronic liver disease to improve the clinical data related to chronic liver disease in China. This cohort study will help us to better manage patients with chronic liver disease and build on this foundation for epidemiology, interventions, and prognosis of chronic liver disease. The cohort and experience generated from this study serves as a support for a series of future studies to focus on clinical issues such as low-level viremia, other complications of cirrhosis, liver failure, end-stage liver disease, and liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who regularly visit and follow up at the corresponding liver disease center
2. All patients meet at least one of the following diagnostic criteria for chronic liver disease:

   * Chronic viral hepatitis B

     * Chronic viral hepatitis C ③. Chronic viral hepatitis D ④. Autoimmune liver disease (PBC/AIH/PSC) ⑤. Non-alcoholic fatty liver disease ⑥. Alcoholic liver disease

Exclusion Criteria:

1. First visit diagnosed with hepatocellular carcinoma or after liver transplantation.
2. Combined with other advanced malignant tumors.
3. The patient refused to sign the informed consent form to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Long-term follow-up of patients with chronic liver disease managed by liver disease centers and infectious disease centers in Shaanxi, Ningxia, Gansu, Qinghai, Xinjiang and other places
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality (liver transplantation) rate in patients with chronic liver disease | 10years
  Clinical data from patients with chronic liver disease are recorded until the patient's death or liver transplantation
Incidence of liver cancer or decompensated cirrhosis in patients with chronic liver disease | 10years
  The incidence of progression to liver cancer or decompensated cirrhosis in patients with chronic liver disease was statistically collected

SECONDARY OUTCOMES:
Incidence of complications related to cirrhosis | 10years
  Incidence of various cirrhosis related complications, including infection, hepatic encephalopathy, gastrointestinal bleeding, ascites, hepatorenal syndrome, etc
Progression rate of liver fibrosis | 10years
  The rate of liver fibrosis progression was assessed by liver tissue biopsy results, fibro scan results, FIB-4 score, APRI score, etc

CONTACTS AND LOCATIONS:
Overall Officials: Yingli He, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital Xi'an Jiaotong University, Xi'an, China